CLINICAL TRIAL: NCT01598688
Title: Monitoring of Cyclosporine Serum Levels in Hematopoietic Stem Cell Transplantation
Brief Title: Cyclosporine (CSA) Level in Blood Samples Collected From Different Lines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Livia Maria Garbin, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CSADOC
Record Dates: First submitted 2012-05-07; First posted 2012-05-15 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Bone marrow transplantation; Hematopoietic stem cell transplantation; Medication management; Nursing care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blood collection immediately after interrupting the drug (Active Comparator): Blood samples were collected from the peripheral venous access, from the catheter line used to infuse the drug and from the line not used for infusion immediately after interrupting the drug infusion.
  Interventions: Other: Blood collection immediately after interrupting CSA infusion
- Blood collection five minutes after interrupting the drug (Experimental): Blood samples were collected from the peripheral venous access, from the catheter line used to infuse the drug and from the line not used for infusion five minutes after interrupting the drug infusion.
  Interventions: Other: Blood collection five minutes after interrupting CSA infusion

INTERVENTIONS:
Other: Blood collection immediately after interrupting CSA infusion — Blood samples were collected from the peripheral venous access, from the catheter line used to infuse the drug and from the line not used for infusion immediately after interrupting the drug infusion.
  For peripheral blood collection, venous access will be established with a small gauge needle.
  The discard method will be adopted for catheter lines collection. Each catheter line is washed with 20 ml of 0.9% normal saline solution, 5 mL of blood are collected and discarded. Using another syringe, the blood volume needed to perform the analysis will then be collected. Additionally, another blood sample will be collected from the catheter line not used to infuse the drug after the discard of 10 mL.
  Other Names: Immediate collection
  Arms: Blood collection immediately after interrupting the drug
Other: Blood collection five minutes after interrupting CSA infusion — Blood samples were collected from the peripheral venous access, from the catheter line used to infuse the drug and from the line not used for infusion five minutes after interrupting the drug infusion.
  For peripheral blood collection, venous access will be established with a small gauge needle.
  The discard method will be adopted for catheter lines collection. Each catheter line is washed with 20 ml of 0.9% normal saline solution, 5 mL of blood are collected and discarded. Using another syringe, the blood volume needed to perform the analysis will then be collected. Additionally, another blood sample will be collected from the catheter line not used to infuse the drug after the discard of 10 mL.
  Other Names: Five minutes
  Arms: Blood collection five minutes after interrupting the drug

SUMMARY:
The purpose of this study is to verify whether differences exist in cyclosporine levels between the samples collected through peripheral venous access, the catheter line used to infuse the drug and the line not used for infusion immediately after interrupting the drug infusion or five minutes after the interruption.

DETAILED DESCRIPTION:
Cyclosporine is an immunosuppressant that prevents graft-versus-host disease, has a narrow therapeutic window, and causes nephrotoxicity. For cyclosporine infusion, a tunneled central venous access device is used; however due to the lipophilic properties of the drug, it can adsorb to the catheter surface and falsely raise cyclosporine concentrations in blood specimens. Some authors recommend sample collection through peripheral access only. Others, however, have shown that these can be collected through the catheter line not used to infuse the drug. Controversies still exist, though, regarding the best timing and blood volume to be discarded to collect the sample.

The hypothesis adopted was that drug adsorption occurs in the line used for infusion. Therefore, there is no statistical or clinical difference between the blood sample collected from the peripheral venous access and from the line not used for cyclosporine infusion. Additionally, this difference becomes smaller when waits five minutes between the interruption of the infusion of the drug and the collection of the blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age who are receiving an allogeneic hematopoietic stem cell transplantation;
* Have a tunneled central venous access device with at least two lines implanted;
* Received cyclosporine administration through this device.

Exclusion Criteria:

* Patients who received cyclosporine infusion through a catheter line other than the one established for this goal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cyclosporine levels in blood samples | At 1 day after the start of the infusion of the drug, and after every seven days during the period the patient is receiving intravenous infusion, an expected average of 4 weeks.

SECONDARY OUTCOMES:
Renal function | Daily since the start of the infusion of the drug, during the period the patient is receiving intravenous infusion, an expected average of 4 weeks.
Liver function | Daily since the start of the infusion of the drug, during the period the patient is receiving intravenous infusion, an expected average of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Livia M Garbin, RN, Principal Investigator — University of Sao Paulo at Ribeirão Preto College of Nursing; Emilia C Carvalho, RN, PhD, Study Director — University of Sao Paulo at Ribeirão Preto College of Nursing
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil